CLINICAL TRIAL: NCT02941874
Title: Determining of Normal Values and Conformity Assessment of the Dosage of a Plasmatic Specific Marker of the Cellular Captation of Glucose: the IRAP Protein (Insulin Regulated AminoPeptidase)
Brief Title: Determining of Normal Values and Conformity Assessment of the Dosage of a Plasmatic Marker of the Cellular Captation of Glucose: the IRAP Protein
Acronym: IRAP
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC16.131
Record Dates: First submitted 2016-10-17; First posted 2016-10-21 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Insulin Resistance
Keywords: IRAP; Insulin Regulated Amino Peptidase; Diagnostic biomarker; Type 2 diabetes
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy volunteers IRAP measurement
  Interventions: Other: Blood sample collection during an OGTT to assess IRAP blood concentration

INTERVENTIONS:
Other: Blood sample collection during an OGTT to assess IRAP blood concentration — Blood sample collection during an OGTT to assess IRAP blood concentration. Blood samples will be collected every 15 minutes during 3 hours

SUMMARY:
The purpose of this study is on one hand to verify the measurement conformity of the IRAP dosage and on the other hand to obtain normal values of the blood IRAP concentration on healthy volunteers.

DETAILED DESCRIPTION:
This study consists of two visits, from two to five days apart.

The first visit :

* Healthy volunteers will be on an empty stomach.
* they will have a clinical examination, blood tests and blood samples will be taken to constitute a blood collection. the IRAP concentration will be measured with those samples.

The second visit : This visit will take place in an interval from 2 to 5 days after the first visit.

* Subjects will be on an empty stomach
* An oral glucose tolerance test (OGTT) of 3 hours will be performed. Blood samples will be taken three time 15 minutes apart at Baseline (before taking the glucose). And then after the glucose intake, blood sample will be taken every 15 minutes to measure insulinemia, blood glucose, and IRAP concentration.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 19 and 25 Kg/m²
* No intercurrent disease during the last week
* No chronic infectious disease
* No smoker, no alcoholic

Exclusion Criteria:

* history of : thyroid disease, liver or renal disease, endocrine and metabolic disease, cardiovascular disease, lung disease, gastroenterological disorders, psychiatric disease, Epilepsy
* Consumption of narcotic drug
* Blood donation dating less than 2 months
* Pregnancy or breast-feeding, or intent to become pregnant during the study period
* legal exclusion criteria

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects distributed according to 3 age groups (40-49 years old , 50-59 years old, 60-70 years old). Every age bracket will be balanced in sex.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Normal values of IRAP concentration will be calculated by making the average of the three dosages of IRAP measured at base line. | At the beginning of the second visit of the study, before the glucose intake
  Three blood samples will be taken 15 minutes apart, before the OGTT. The average of IRAP concentration measured with those 3 samples, will be used to assess the normal values of IRAP concentration on a healthy population.

SECONDARY OUTCOMES:
Repeatability of the IRAP measurement | At the beginning of the second visit of the study, before the glucose intake
  The repeatability will be assessed during the second visit. The measurement of IRAP concentration will be repeated 3 times on the first sample taken before the OGTT.
Temporal reproducibility of the concentration of IRAP | At the beginning of the second visit of the study, before the glucose intake
  The reproducibility will be assessed during the second visit. The measurement of IRAP concentration will be repeated 3 times on the first sample taken before the OGTT.

OTHER OUTCOMES:
kinetic profile of the concentration of IRAP during OGTT | During the 3 hours OGTT at the second visit
  Evolution of the serum concentration of IRAP during the 3 hours which follow the ingestion of 75g of glucose.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Biologie - Pathologie, Grenoble, Isere, France